CLINICAL TRIAL: NCT03401021
Title: Factors Associated With Quit Intention Among Male Smokers Whose Partner Got Pregnant: An Exploration Study
Brief Title: Factors Related to the Intention to Quit Among Male Smokers During Their Wives Pregnancy
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW17-509
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Smoking Cessation
Keywords: intention to quit smoking; male smoker; smoking cessation; expectant fathers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crrent Male smokers: Male smokers met the inclusion criteria below will be invited to fill in the questionnaires set, part of them will be invited to attend a semi-structured interview(optional).
  1. be aged 18 or above,
  2. have a history of smoking at least one cigarette per day before their partners became pregnant,
  3. be involved with partners whose pregnancies could be confirmed,
  4. able to read Chinese and communicate in the Mandarin dialect.
  Interventions: Other: Questionnaires set

INTERVENTIONS:
Other: Questionnaires set — Participants will be asked to respond to the demographic information sheet, Smoking characteristics sheet, the Fagerstrom Test of Nicotine Dependence, the Transtheoretical Model (TTM) variables, Smoking Self-efficacy Questionnaire (SEQ-12), Family Adaptation, Partnership, Growth, Affection, and Resolve (Family APGAR), and a smoking hazard questionnaire.

SUMMARY:
This study aims to use a cross-sectional study and semi-structured interview to explore the level of intention to quit smoking among male smokers whose partner got pregnant and further explore factors associated with their quit intention.

DETAILED DESCRIPTION:
With a globally growing number of smokers, up to about half of men and one tenth of women are becoming smokers and relatively few stopping, especially in Mainland China.

It has been proved that tobacco is responsible for even more deaths and diseases. Smokers have two to three times mortality in middle age among otherwise similar persons who had never smoked. According to the literature review, smoking has been confirmed to be an important risk factor to coronary heart disease, chronic obstructive lung disease, cancer, stroke, peptic ulcer, peripheral vascular disease, and so on. In addition, tobacco can also increase the incidence rate of cancer in lung, oral cavity, naso-, oro- and hypopharynx, nasal cavity et.al, as well as myeloid leukemia, among smokers.

For the male smokers at their reproductive ages, who is preparing to have a baby with their partners, smoking may negatively influence their reproductive capacity. Sufficient studies found that the quantity and duration of smoking, especially the current smoking is positively associated with the risk of erectile dysfunction. Smoking may increase the risk of a higher risk of developing oligospermia, asthenozoospermia and teratozoospermia for man in the reproductive years, which may lead to the inefficiency of fertilization and even give birth to abnormal fetus. Besides, secondhand Smoking (SHS) exposure also have further and longer negative effects on their female partner and their baby born in the future. The non-smoking population is much more sensitive to the nicotine in the passive smoking than smokers. The SHS may increase the risk of respiratory infections, ear problem, immediate adverse effects on cardiovascular system, CHD, lung cancer and so on to adults. For the children, the passive smoking makes children have a higher chance to get severe asthma, slow lung growth. Hence, children and women live with smokers may have a higher risk of premature death and disease. Besides, newborns whose mothers were exposed to secondhand smoking showed significantly lower scores in the habituation cluster and motor system cluster [16], as well as the delay of neurobehavioral development regardless of socio-demographic, obstetric and pediatric factors. Conclusively, smoking has direct and indirect negative effect to male smokers in reproductive ages themselves and their family members.

Based on the official statistic figures in 2010, about one third of people in China were current smokers, and the number of young smokers is increasing [4]. While most current smokers (83.9%) report having no intention to quit smoking (WHO, 2011). On average, between 60% and 70% of Chinese men continue to smoke into middle age, which is different with the western countries. Hence, finding out a solution to decrease the married reproductive male smoking rate is extremely crucial.

Overall awareness of the health hazards of tobacco has improved in the last 15 years in China, but is still relatively poor. Even there were several patterns of propaganda and education applied in China, the efficiency is not very satisfactory. Hence, an effective education intervention that delivery the health hazards of tobacco to male smokers and secondhand smoking to their wives and baby born in the future should be developed and implemented for reproductive male smokers in China.

Cigarette can negatively influence the function of respiratory, urinary and other systems, as well as increase the risk of different types of cancer. Secondhand smoking is harmful to their family members. What's worse, the impact of the reproductive system will further damage their baby born in the future. As the overlooking of the impact of maternal smoking on the fetus, the smoking cessation research for the male smokers who plan to have a baby is absent. For Chinese people, the high prevalence and low quitting rate made this situation much worse. In addition, as the cancel of the one-child policy, lots of couples are planning to give birth to a baby in the future decades compared with the period the policy was valid. Considering the high prevalence of male smoking and upcoming high birth rate in China, more smokers, pregnant, and fetus are under the hazard of tobacco use.

Before applying interventions to help male smokers whose partner got pregnant to quit or reduce cigarette smoking, a study exploring their intention to quit smoking and relevant factors must be implemented.

ELIGIBILITY:
Inclusion Criteria:

* (1) All participants should be males
* (2) All participants should be aged 18 or above;
* (3) All participants should be married;
* (4) All participants should be smoking at least one cigarette per day averagely during the past 3 months;
* (5) All participants should be able to communicate in Mandarin (including reading Chinese)

Exclusion Criteria:

* Smokers who meet the above criteria but are currently involved in other smoking cessation programs or the pilot study and/or mentally or physically unfit for communication will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the participant eligibility is based on both biological and self-representation of gender identity, smokers who is male biologically and also reported as a male will be eligible in this study.
Study Population: The study population is include males smokers who is/will planning to have a baby with their partners.
Sampling Method: Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Quit intention of smoking | Baseline
  The level of intention to quit of smoking among male smokers who planning to have a baby with their partners will be measured by b) The Transtheoretical Model (TTM) variables. The Stage of TTM will be assessed by asking the intention of quitting smoking in the past 6 months with the 6-items, which are Precontemplation, Contemplation, Preparation, Action, Maintenance, and Termination

SECONDARY OUTCOMES:
Self-efficacy level | Baseline
  Self-efficacy of participants against tobacco will be assessed by using by the SEQ-12. The SEQ-12 is categorized into two subscales, namely internal stimuli (6 items) and external stimuli (6 items), with total possible scores ranging from 6 to 30 for both internal stimuli and external stimuli. Higher scores of the SEQ-12 on both subscales indicate greater self-efficacy to refrain from smoking.
Self-awareness of the hazard of smoking | Baseline
  The self-awareness of the hazard of smoking among the participants will be measured by a self-designed smoking hazard questionnaire list. The smoking hazard questionnaire lists 14 hazard of smoking and SHS to the pregnant, fetus, health, income, social activity, and so on. Participants responded to each items using a -10 to 10 rating scale ranging from -10 (most negative influence) to 10 (most positive influence).
Family support level | Baseline
  The family support for smoking cessation will be assessed by using the Family APGAR. The Family APGAR is a 5-item measure of perceived family support [71]. Participants responded to each item using a 5-point rating scale ranging from 0 (never) to 4 (always). The standard scoring for the FAPGAR interprets high scores (7-10) as indicating a satisfactory support from family and low scores (0-3) indicating severe dysfunctionality support from the family members.
Dependence of nicotine | Baseline
  The level of nicotine dependence of the participants will be measured by the Fagerstrom Test of Nicotine Dependence (FTND) scale. The FTND is a standard instrument for assessing the intensity of physical addiction to nicotine.The test was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerstrom score, the more intense is the patient's physical dependence on nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia W, Li HCW, Song P, Ho KY, Luo Y, Liang T, Ho LLK, Cheung AT, Cai W. Perceptions, behaviours and attitudes towards smoking held by the male partners of Chinese pregnant women: a qualitative study. BMC Public Health. 2021 Oct 20;21(1):1901. doi: 10.1186/s12889-021-11966-4. PMID 34670560